CLINICAL TRIAL: NCT02630979
Title: Prospective Observational Questionnaire Based Study Measuring Oncology Physicians Knowledge and Satisfaction With the Outcomes of Expensive Cytotoxic Agents
Brief Title: Oncologists Satisfaction With Outcomes of Some Cytotoxic Agents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mahmoud Ellithy, Associate professor of clinical oncology. Ain Shams University, Ain Shams University
Other Study IDs: Cure and more1
Record Dates: First submitted 2015-12-06; First posted 2015-12-15 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2016-05

CONDITIONS: Physician Satisfaction With the Outcomes of Cytotoxic Drugs
MeSH Terms: interventions — Bias

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — No biospecimen
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment: Clinical and medical oncology physicians.
  Interventions: Behavioral: Measuring satisfaction, knowledge and bias

INTERVENTIONS:
Behavioral: Measuring satisfaction, knowledge and bias — Questionnaire based assessment.

SUMMARY:
The study measures the degree of oncology physician satisfaction with the outcomes of some cytotoxic agents.

DETAILED DESCRIPTION:
This is a prospective observational questionnaire based study measuring the degree of satisfaction of medical oncologists with the results of some expensive cytotoxic agents. The study also measures the physician knowledge with the toxicity profile of the tested drugs, pharmaceutical perspectives, methods of administration, adherence to guidelines and the degree of bias of the physicians when prescribing this drugs.

The tested drugs are trastuzumab, lapatinib, sunitinib, m tor inhibitors, sorafenib, cetuximab, panitumumab, bevacizumab, erlotinib, rituximab, imatinib mesylate, gefitinib, abiraterone acetate, cabazitaxel, pertuzumab, fulvestrant, pemetrexate and crizotinib.

The evaluation will be through a predesigned questionnaire ( 30 questions ). The questions are divided into four categories measuring four items, the degree of physician satisfaction with the drugs results and toxicity profile, orientation with pharmaceutical perspectives of the drugs, adherence to guidelines and degree of bias with pharmaceutical companies complements. A predesigned questionnaire based scoring system will categorise the processed data to low, intermediate and high score for each of the four measured topics. The data will be processed and the degree of satisfaction, orientation with pharmaceutical perspectives, adherence to guidelines and degree of bias will be grade to low, moderate or high. Subsequent recommendations for cost effective analysis, physician education and strict auditing measures for drug prescription will be elaborated for the drugs.

NB: The study will be on two waves. The first wave will evaluate 9 drugs and the second wave will evaluate 8 drugs.

ELIGIBILITY:
Inclusion Criteria:

* Physicians ranked from senior resident to professional consultants

Exclusion Criteria:

* Junior residents.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical or clinical oncology doctors
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Questionnaire based measurement of the degree of physician satisfaction with the results and toxicity of some cytotoxic drugs. | One year
  A predesigned questionnaire based scoring system will categorise the degree of satisfaction to low, intermediate and high score.
Questionnaire based measurement of the degree of physician orientation with pharmaceutical perspectives of some cytotoxic drugs. | One year
  A predesigned questionnaire based scoring system will categorise the degree of orientation to low, intermediate and high score.
Questionnaire based measurement of the degree of physician adherence to guidelines in prescribing some cytotoxic drugs. | One year
  A predesigned questionnaire based scoring system will categorise the degree of adherence to guidelines to low, intermediate and high score.
Questionnaire based measurement of the degree of physician bias while prescribing some cytotoxic drugs. | One year
  A predesigned questionnaire based scoring system will categorise the degree of bias to low, intermediate and high score.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Ellithy, Consultant, Principal Investigator — Faculty of Medicine. Ain Shams University; Noha Salaheldin elbogdady, Pharmaciest, Study Director — Misr university
Locations (1):
- Faculty of Medicine. AIn Shams University, Cairo, Elabbasia, Egypt

IPD SHARING:
Plan to Share IPD: Yes